CLINICAL TRIAL: NCT04431583
Title: Transition of Single Surgeon Bariatric Service to an Interdisciplinary Multiple Surgeon Model
Status: Completed | Type: Observational
Sponsor: University of Adelaide (Other)
Collaborators: Central Adelaide Local Health Network Incorporated (Other Government)
Responsible Party: Principal Investigator, Antonio Barbaro, Associate Clinical Lecturer, University of Adelaide
Other Study IDs: 13204
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 2008-2012 Participants: Participants who underwent bariatric surgery between 2008 and 2012 (inclusive).
  Interventions: Procedure: Bariatric surgery- single surgeon service
- 2013-2016 Participants: Participants who underwent bariatric surgery between 2013 and 2016 (inclusive).
  Interventions: Procedure: Bariatric surgery- multiple surgeon + multidisciplinary team approach
- 2017- 2018 Participants: Participants who underwent bariatric surgery between 2017 and 2018 (inclusive).
  Interventions: Procedure: Bariatric surgery: formalized streamlined multiple surgeon + multidisciplinary team approach

INTERVENTIONS:
Procedure: Bariatric surgery- single surgeon service
  Groups: 2008-2012 Participants
Procedure: Bariatric surgery- multiple surgeon + multidisciplinary team approach
  Groups: 2013-2016 Participants
Procedure: Bariatric surgery: formalized streamlined multiple surgeon + multidisciplinary team approach
  Groups: 2017- 2018 Participants

SUMMARY:
This retrospective study will analyse the transition of an Australian hospital which significantly increased volume of bariatric operations after introduction of a clinical pathway, and to assess the outcomes. Barriers to introduction of the multidisciplinary pathway and the means to overcome these will also be analysed and discussed. The analysis will also determine if there are any other areas of bariatric surgery which can be further investigated to optimise current practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have had bariatric surgery at The Queen Elizabeth Hospital between 2008-2018

Exclusion Criteria:

* nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent bariatric surgery at the Queen Elizabeth Hospital (South Australia) between the years of 2008 and 2018.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Post-operative length of stay (nights) | The number of nights the participant stay in hospital from the day of procedure to the day of hospital discharge. This time period occurs immediately after the procedure. This data will be retrospectively reviewed on an average of 5 years.
  This will be measured in number of nights the participant stayed in hospital after the procedure.
End weight loss | Up to 12 months
  Post-operative weight loss

SECONDARY OUTCOMES:
End weight loss | Up to 24 months
  Post-operative weight loss
End weight loss | Up to 36 months
  Post-operative weight loss
Intraoperative time | The start time of the operation to the end time of the procedure. This data will be retrospectively reviewed on an average of 5 years.
  Duration of operative time measured in minutes
Post-operative complications | Up to 36 months
  Complications which occurred in the post operative period
Number of operations performed in time period | Retrospectively reviewed, 1 yearly
  The number of operations which occurred in each group
Type of Operation Performed | Retrospectively reviewed, 1 yearly
  The number of the different types of bariatric operations which occurred in each group
Number of participants converted from Gastric Sleeve to Gastric Bypass | Retrospectively reviewed, 1 yearly
Number of patients on surgical waitlist | Retrospectively reviewed, 1 yearly
  The number of patients on the surgical waitlist for each time period

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Barbaro, MBBS, Principal Investigator — University of Adelaide; Harsh Kanhere, MS, FRACS, AFRACMA, Study Director — Central Adelaide Local Health Network; Markus Trochsler, MD, FMH, MMIS, FRACS, Study Director — Central Adelaide Local Health Network; Gayatri Asokan, MBBS, FRACS, Principal Investigator — Central Adelaide Local Health Network; Matheesha Herath, MBBS, Principal Investigator — Central Adelaide Local Health Network; Raghav Goel, MBBS, Principal Investigator — Central Adelaide Local Health Network

IPD SHARING:
Plan to Share IPD: No